CLINICAL TRIAL: NCT02585700
Title: A Phase 1 Double Blinded, Randomized, Placebo-Controlled Study to Examine the Safety and Immunogenicity of a Seasonal Trivalent Split, Inactivated Influenza Vaccine Produced by Torlak in Healthy Adult Volunteers in Serbia
Brief Title: A Study of a Seasonal Trivalent Split, Inactivated Influenza Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Virology, Vaccines and Sera, Torlak (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); World Health Organization (Other); PATH (Other); Comac Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TORLAK-100
Record Dates: First submitted 2015-10-13; First posted 2015-10-23 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2015-10

CONDITIONS: Influenza, Human
Keywords: Grippe; Human Flu; Human influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine (Experimental): 0.5 mL of influenza vaccine, split, inactivated with 15 mcg of haemagglutination (HA) of each of 3 strains:
  * NYMC BX-51B reassortant of B/Massachusetts/2/2012
  * X-181 reassortant of H1/A/California/7/2009
  * X-223A reassortant of H3/A/Texas/50/2012.
  Interventions: Biological: Influenza vaccine, split inactivated
- Placebo (Placebo Comparator): 0.5 mL of phosphate buffered saline
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Influenza vaccine, split inactivated — Seasonal trivalent inactivated influenza vaccine (TIV), inactivated split virion, purified by sucrose gradient ultracentrifugation. The vaccine is produced in hen's eggs, and inactivated with beta-propiolactone.
  Arms: Vaccine
Other: Placebo — 0.5 mL of phosphate buffered saline
  Arms: Placebo

SUMMARY:
This is a phase I, double-blind, randomized, placebo-controlled trial with two groups of participants to receive seasonal trivalent split, inactivated influenza vaccine (A/H1N1; A/H3N2 and B) or placebo (phosphate buffered saline). A total of 60 healthy male and female adults 18 through 45 years of age will be randomized to receive vaccine (30) or placebo (30).

DETAILED DESCRIPTION:
This is a phase 1, double blinded, randomized, placebo-controlled study. The study will be conducted at 1 site in Serbia. Sixty (60) healthy male and female adults, 18 to 45 years of age, will be enrolled into the trial. Subjects will be randomized 1:1 to one of two treatment allocations: 30 to vaccine, 30 to placebo. The study will utilize a "randomized block design" to assure a balance of 1:1 vaccine and placebo when all subjects are enrolled. The study will be double blinded, meaning the study subjects, investigators, and the sponsor will be unaware of the treatment allocated to each subject until the clinical trial database is declared final and locked. The study should take about 5 months to complete, with each subject involved for 3 months from the day of injection. The justification for the 3 month follow up, rather than 6 month follow up is that this is an inactivated vaccine that follows very standard manufacturing practices with standard antigens. The safety of inactivated influenza vaccines is well-established. Adding length to the follow up results in delays in future testing of the vaccine for licensure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adult 18 through 45 years of age at the enrollment visit.
* Literate (by self-report) and willing to provide written informed consent.
* Healthy, as established by the medical history, physical examination, and screening laboratory evaluations.
* Capable and willing to complete Memory Aids and willing to return for all follow-up visits.
* For females, willing to utilize reliable birth control measures (e.g., intrauterine device, hormonal contraception, condoms) from Day 0 through the Day 21 visit.

Exclusion Criteria:

* Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during the period of this study.
* Receipt of any non-study vaccine within 4 weeks prior to enrollment or refusal to postpone receipt of such vaccines until after the Day 21 visit.
* Current or recent (within 2 weeks of vaccination) acute illness with or without fever.
* Receipt of immune globulin or other blood products within 3 months prior to study enrollment or planned receipt of such products prior to the Day 21 visit.
* Chronic administration (defined as more than 14 consecutively-prescribed days) of immunosuppressants or other immune-modulating therapy within six months prior to study vaccination. (For corticosteroids, this means prednisone or equivalent, equal or more than 0.5 mg per kg per day; topical steroids are allowed.)
* History of asthma.
* Hypersensitivity after previous administration of any vaccine.
* Suspected or known hypersensitivity to any of the study vaccine components, including chicken or egg protein.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatobiliary, metabolic, neurologic, psychiatric or renal functional abnormality, as determined by medical history, physical examination or clinical laboratory screening tests, which in the opinion of the investigator, might interfere with the study objectives.
* History of any blood or solid organ cancer.
* History of thrombocytopenic purpura or known bleeding disorder.
* History of seizures.
* Known or suspected immunosuppressed or immunodeficient condition of any kind.
* Confirmed hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Known HIV infection (self-report).
* Known active tuberculosis or symptoms of active tuberculosis, regardless of cause (self-report).
* History of chronic alcohol abuse and/or illegal drug use.
* Pregnancy or lactation. (A negative pregnancy test will be required before administration of study product for all women of childbearing potential.)
* History of Guillain-Barré Syndrome
* Any condition that, in the opinion of the investigator, would increase the health risk to the subject if he/she participates in the study or would interfere with the evaluation of the study objectives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Goran Stevanovic, PhD, Principal Investigator — Clinic for Infectious and Tropical Diseases
Locations (1):
- Clinical Center of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stevanovic G, Lavadinovic L, Filipovic Vignjevic S, Holt R, Ilic K, Berlanda Scorza F, Sparrow E, Stoiljkovic V, Torelli G, Madenwald T, Socquet M, Barac A, Ilieva-Borisova Y, Pelemis M, Flores J. Safety and immunogenicity of a seasonal trivalent inactivated split influenza vaccine: a phase I randomized clinical trial in healthy Serbian adults. Hum Vaccin Immunother. 2018 Mar 4;14(3):579-586. doi: 10.1080/21645515.2017.1415683. Epub 2018 Feb 23. PMID 29239682

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All volunteers were recruited at the Clinical Center of Serbia, Belgrade, Serbia.
Pre-assignment Details: 66 people were screened for the study after signing consent. 6 subjects failed screening. A total of 60 subjects received vaccine or placebo.
Groups:
- Vaccine Group: 0.5 mL of influenza vaccine split, inactivated with 15 mcg of HA of B/Massachusetts, H1/A/California, and H3/A/Texas
- Placebo Group: 0.5 mL of phosphate buffered saline
Period: Overall Study
Arm/Group | Vaccine Group | Placebo Group
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine Group | Placebo Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.00 (7.21) | 30.70 (6.14) | 30.85 (6.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 21 | 21 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 30 | 30 | 60
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Serbia | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Immediate Adverse Events
Description: Number of subjects with observed immediate adverse events, including allergic reaction or anaphylaxis, following administration of the study product.
Time Frame: 30-minute post-vaccination period.
Population: The analysis was conducted for subjects who were randomized and received a study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

2. Primary Outcome: Number and Percentage of Subjects With Solicited Local Reactogenicity
Description: Number of subjects reporting solicited local reactions (redness, swelling, induration, pain and tenderness) at the injection site post-vaccination with study vaccine or placebo
Time Frame: 7-day period (Days 0-6) post-vaccination.
Population: The analysis was conducted for subjects who were randomized and received a study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Participants
  Hardness | 2 | 0
  Pain | 14 | 4
  Redness | 6 | 0
  Swelling | 2 | 0
  Tenderness | 10 | 1

3. Primary Outcome: Number and Percentage of Subjects With Solicited Systemic Reactogenicity
Description: Number of subjects reporting solicited systemic reactions (fever, fatigue/malaise, muscle aches, joint aches, chills, nausea, vomiting, and headache) post-vaccination with study vaccine or Placebo
Time Frame: 7-day period (Days 0-6) post-vaccination.
Population: The analysis was conducted for subjects who were randomized and received a study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Participants
  Temperature above 37 C | 2 | 1
  Chills | 2 | 0
  Headache | 5 | 2
  Joint aches | 1 | 2
  Muscle aches | 2 | 1
  Nausea | 2 | 0
  Tiredness | 5 | 0
  Vomiting | 1 | 0

4. Primary Outcome: Number and Percentage of Subjects With Occurrence of Unsolicited Adverse Events
Description: These data are presented broadly as number per group for the study. Please see AE reporting section for more specific details on AEs.
Time Frame: Within 21 days post vaccination
Population: The analysis was conducted for subjects who were randomized and received a study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Participants | 2 | 4

5. Primary Outcome: Number and Percentage of Subjects With Occurrence of Serious Adverse Events (SAE)
Time Frame: Over the entire study period (Day 90).
Population: The analysis was conducted for subjects who were randomized and received a study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Participants
  Serious adverse events (SAEs)--related | 0 | 0
  SAEs--not related | 0 | 0

6. Secondary Outcome: Number and Percentage of Seroconverted Subjects Against 3 Strains of Influenza Vaccine.
Description: Seroconversion is defined as a serum HAI titer meeting the following criteria:
  * pre-vaccination titer <1:10 and a post-vaccination titer ≥ 1:40 or
  * pre-vaccination titer ≥ 1:10 and at least a four-fold increase in post-vaccination measured on Day 21.
  The 3 influenza strains assessed were B/Massachusetts, H1/A/California and H3/A/Texas
Time Frame: Day 21
Population: The analysis was conducted for subjects who were randomized and received a study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Participants
  Seroconversion to H1 | 25 | 0
  Seroconversion to H3 | 23 | 0
  Seroconversion to B | 21 | 0

7. Secondary Outcome: Number and Percentage of Seroprotected Subjects Against 3 Strains of Influenza Vaccine
Description: A seroprotected subject was defined as a vaccinated subject who had a serum Hemagluttination Inhibition (HAI) titer ≥ 1:40. The 3 influenza strains assessed were B/Massachusetts, H1/A/California an d H3/A/Texas
Time Frame: Day 0 and Day 21 post vaccination
Population: All vaccinated subjects who have valid post vaccination immunogenicity measures with no major protocol violations
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Participants
  H1 | 30 | 10
  H3 | 30 | 19
  B | 26 | 5

8. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Antibodies Pre- (Day 0) and Post-vaccination (Day 21) for Each of the 3 Antigens
Description: The 3 influenza strains assessed were B/Massachusetts, H1/A/California an d H3/A/Texas
Time Frame: Pre- (Day 0) and post-vaccination (Day 21)
Population: All vaccinated subjects with no major protocol violations who have valid post vaccination immunogenicity measures
Measure: Mean (95% Confidence Interval); unit: Titers
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Titers
  GMT to H1 Day 0 | 15.97 [11.30 to 23.10] | 21.19 [14.82 to 30.29]
  GMT to H1 Day 21 | 295.14 [240.10 to 362.80] | 22.32 [15.72 to 31.69]
  GMT to H3 Day 0 | 37.75 [25.88 to 55.07] | 41.41 [28.02 to 61.20]
  GMT to H3 Day 21 | 439.67 [320.54 to 603.06] | 42.87 [28.92 to 63.55]
  GMT to B Day 0 | 10.47 [7.91 to 13.86] | 10.72 [7.72 to 14.89]
  GMT to B Day 21 | 75.95 [56.88 to 101.40] | 10.66 [7.69 to 14.76]

9. Secondary Outcome: Geometric Mean Fold Rises (GMFRs) of Serum (HAI) Antibodies (Post-vaccination / Pre-vaccination) for Each of the 3 Antigens.
Description: The 3 influenza strains assessed were B/Massachusetts, H1/A/California an d H3/A/Texas
Time Frame: Pre- (Day 0) and post-vaccination (Day 21)
Population: All vaccinated subjects who have valid post vaccination immunogenicity measures with no major protocol violations
Measure: Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
fold rise
  GMFR for H1 | 18.49 [12.22 to 27.95] | 1.05 [1.00 to 1.11]
  GMFR for H3 | 11.65 [7.82 to 17.35] | 1.04 [.99 to 1.08]
  GMFR for B | 7.25 [5.53 to 9.52] | 0.99 [.96 to 1.03]

10. Secondary Outcome: Geometric Mean Neutralization Titers of Neutralizing Antibodies (MNT) Pre- (Day 0) and Post-vaccination (Day 21) for Each of the 3 Antigens.
Time Frame: Pre- (Day 0) and post-vaccination (Day 21)
Population: All vaccinated subjects who have valid post vaccination immunogenicity measures with no major protocol violations
Measure: Mean (95% Confidence Interval); unit: Titers
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
Titers
  GMT to H1 Day 0 | 24.06 [18.61 to 31.11] | 31.75 [24.06 to 41.89]
  GMT to H1 Day 21 | 211.12 [164.95 to 270.22] | 40.00 [30.47 to 52.52]
  GMT to H3 Day 0 | 18.02 [12.74 to 25.51] | 19.77 [15.11 to 25.86]
  GMT to H3 Day 21 | 125.53 [87.82 to 179.45] | 24.34 [18.39 to 32.22]
  GMT to B Day 0 | 80.93 [59.21 to 110.61] | 70.45 [48.06 to 103.28]
  GMT to B Day 21 | 331.28 [278.78 to 393.68] | 105.56 [75.73 to 147.15]

11. Secondary Outcome: Geometric Mean Fold Rises (GMFRs) of MNT (Post-vaccination / Pre-vaccination) for Each of the 3 Antigens.
Description: The 3 influenza strains assessed were B/Massachusetts, H1/A/California an d H3/A/Texas
Time Frame: Pre- (Day 0) and post-vaccination (Day 21)
Population: All vaccinated subjects who have valid post vaccination immunogenicity measures with no major protocol violations
Measure: Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 30 | 30
fold rise
  GMFR for H1 | 8.77 [6.70 to 11.49] | 1.26 [1.09 to 1.45]
  GMFR for H3 | 6.96 [4.89 to 9.92] | 1.23 [1.14 to 1.33]
  GMFR for B | 4.09 [3.11 to 5.38] | 1.50 [1.18 to 1.89]

ADVERSE EVENTS:
Time Frame: 90 days
Groups:
- Vaccine Group: 0.5 mL of influenza vaccine, split, inactivated with 15 mcg of HA of each of 3 strains:
  * NYMC BX-51B reassortant of B/Massachusetts/2/2012
  * X-181 reassortant of H1/A/California/7/2009
  * X-223A reassortant of H3/A/Texas/50/2012.
Arm/Group | Vaccine Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 2/30 | 4/30
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine Group (N=30) | Placebo Group (N=30)
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Unrelated to study product
Diarrhea (Gastrointestinal disorders) | 0 | 1 — Unrelated to study products
Alanine Aminotransferase Increased (Investigations) | 0 | 1 — Unrelated to study products
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 — Unrelated to study products
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Unrelated to study products

LIMITATIONS AND CAVEATS:
No limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No